CLINICAL TRIAL: NCT05051943
Title: A Prospective Observational Study of the Real-world Use of an Adalimumab Biosimilar and Evaluation of Nutritional Status on the Therapeutic Response
Brief Title: A Study of the Real-world Use of an Adalimumab Biosimilar and Evaluation of Nutritional Status on the Therapeutic Response
Acronym: OPALE
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: ADAL-001-CNI
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Crohn Disease; Ulcerative Colitis; Psoriasis; Ankylosing Spondylitis; Rheumatoid Arthritis; Psoriatic Arthritis
Keywords: nutrition
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Psoriasis; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe the real-world profile of patients treated with adalimumab FK in gastroenterology, dermatology or rheumatology in order to evaluate in this population the predictive factors of therapeutic response (in particular nutritional status) and generate hypothesis between nutritional status and therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old who agree to participate in the study and do not object to the use of their health data
* A disorder treated with anti-TNF therapy
* Whose physician made the decision to initiate adalimumab treatment prior to the study

Exclusion Criteria:

* Patients participating in an interventional therapeutic trial at the time of inclusion
* Patients who are unwilling or unable to fulfil follow-up requirements (patients who cannot be reached by phone or complete the self-administered questionnaire or not fluent in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with rhumatologic, gastrologic or dermatologic disease eligible to a treatment with adalimumab
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) | 12 months
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Peyrin-Biroulet, MD, Principal Investigator — CHU NANCY
Locations (1):
- CHRU de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, France